CLINICAL TRIAL: NCT06735495
Title: The Safety and Efficacy of CD19 & CD22 Bispecific CAR T Cells in Treating Relapsed / Refractory B Cell Hematological Tumors
Brief Title: CD19 & CD22 Bispecific CAR T Cells in the Treatment of Relapsed/Refractory B Cell Hematologic Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Hebei Taihe Chunyu Biotechnology Co., Ltd (Industry)
Responsible Party: Principal Investigator, MEI HENG, Proferssor, Cheif Doctor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19 & CD22 bispecific CAR T
Record Dates: First submitted 2024-12-05; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: B-Cell Lymphoblastic Leukemia/Lymphoma
Keywords: CAR-T; dual-target; Relapsed / Refractory B Cell Hematological Tumors
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effective of CD19&CD22 bispecific CAR-T cells (Experimental): The infusion dose range of cells in this trial is recommended: 1 to 2 10^6 And CAR-T cells / kg.
  Interventions: Drug: CD19&CD22 bispecific CAR-T cells

INTERVENTIONS:
Drug: CD19&CD22 bispecific CAR-T cells — Each patient will receive CD19&CD22 bispecific CAR-T cells by intravenous infusion on day 0

SUMMARY:
This study is a multi-center, open, prospective single-arm clinical study of patients with relapsed / refractory B cell hematological tumors to evaluate the safety and efficacy of CD19 & CD22 bispecific CAR-T cells in relapsed / refractory B cell hematological tumors while collecting pharmacokinetics and pharmacodynamics indicators of CAR-T cells.

DETAILED DESCRIPTION:
Since 2010, CAR-T ( chimeric antigen receptor T cell) therapy has shown good results in tumor treatment and has achieved positive clinical therapeutic effects in hematological tumors. The structure of the dual-target CAR-T of CD19 & CD22 is designed with a 4-1BB costimulatory domain and an antigenic recognition region with a tandem structural sequence to recognize CD22 or CD19 by a single structure. CD19 & CD22 bispecific CAR-T cells can identify CD 19 or CD 22 with the advantage that the single target CAR-T does not have, reducing the possibility of target loss. The structure has been optimized to enhance the safety to treat B cell-derived hematological tumors (at least CD19 positive or CD22 positive).

ELIGIBILITY:
Inclusion Criteria:

1.CD 19 + / CD 22 + B cell hematological tumor was confirmed by pathological and histological examination, and the patient met the following criteria for relapsed or refractory B cell hematological tumor:

1. Refractory / relapsed B lymphocytic leukemia (1 of the following 4 items can be met):

   i . Recurrence within 6 months of first remission; ii. Primary refractory without complete remission after 2 cycles of standard chemotherapy regimen; iii. No complete remission or recurrence after first-line or multiline salvage chemotherapy; iv. Not eligible for HSCT conditions, abandonment of HSCT, or relapse after HSCT due to conditional limitations.
2. Refractory / relapsed B-cell lymphoma (meet the following item 1 of the first 4 items plus item 5):

i . After four courses of chemotherapy with a standard regimen, tumor shrinkage was less than 50% or disease progression; ii . CR after standard regimen chemotherapy, but relapsed within 6 months; iii.2 or more recurrences after CR; iv . Not suitable for hematopoietic stem cell transplantation, or abandoning HSCT due to conditional restrictions or relapse after hematopoietic stem cell transplantation; v . Subject must have received prior adequate treatment, including at least: a monoclonal antibody against CD 20 and combination chemotherapy containing an anthracycline drug agent.

2.The results of FCM or immunohistochemical detection of tumor antigen (CD 19 / CD 22) were positive.

3.The estimated survival period is more than 3 months starting from the signing of the informed consent form.

4.Good organ function,Meet the following requirements：

1. HGB≥70g/L(transfusible)
2. Liver and kidney function: creatinine ≤1.5XULN: total bilirubin ≤1.5XULN:ALT and AST≤2.5X ULN
3. Cardiopulmonary function: left ventricular ejection fraction >50%; Blood oxygen saturation >90%;

5.Subjects with the Eastern Cooperative Oncology Group (ECOG) fitness scores of 0 to 2.

Exclusion Criteria：(If meet any of the following criteria, patients will not be included)

1. Serious heart insufficiency,LVEF <50%
2. History of severe pulmonary function impairment disease.
3. Other malignant tumors in the advanced stage.
4. Severe infection or persistent infection that cannot be effectively controlled.
5. Combined with severe autoimmune disease or innate immune deficiency.
6. Active hepatitis (hepatitis B virus deoxyribonucleic acid [HBV-DNA 500 IU / ml and abnormal liver function] or hepatitis C antibody [HCV-Ab] positive, HCV-RNA above the lower limit of detection of the analytical method and abnormal liver function).
7. Human immunodeficiency virus (HIV) infection or syphilis infection.
8. History of severe allergies to biological products (including antibiotics).
9. Acute graft-versus-host response (GVHD) allogeneic hematopoietic stem remained one month after immunosuppressant discontinuation.
10. Patients who have other serious physical or mental illnesses or abnormalities in laboratory tests that may increase the risk of participating in the clinical trial or interfere with the study results, and who are deemed unsuitable for participation in the clinical trial by the investigator

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) of administering CD19&CD22 dual-target CAR-T cells In the treatment of relapsed/refractory B-cell hematologic tumors | within 3 years after infusion
  Disease overall response rate (ORR) will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Complete response rate (CR) of administering CD19&CD22 dual-target CAR-T cells In the treatment of relapsed/refractory B-cell hematologic tumors | within 3 years after infusion
  CR will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Complete response with incomplete blood recovery rate (CRi) of administering CD19&CD22 dual-target CAR-T cells In the treatment of relapsed/refractory B-cell hematologic tumors | within 3 years after infusion
  CRi will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Partial response rate (PR) of administering CD19&CD22 dual-target CAR-T cells In the treatment of relapsed/refractory B-cell hematologic tumors | within 3 years after infusion
  PR will be assessed from CAR-T cell infusion to death or last follow-up.

SECONDARY OUTCOMES:
Duration of Response (DOS) of administering CD19&CD22 dual-target CAR-T cells in the treatment of relapsed/refractory B-cell hematologic tumors | within 3 years after infusion
  DOS will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Progress-free survival (PFS) of administering CD19&CD22 dual-target CAR-T cells in the treatment of relapsed/refractory B-cell hematologic tumors | within 3 years after infusion
  PFS will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Overall survival (OS) of administering CD19&CD22 dual-target CAR-T cells in the treatment of relapsed/refractory B-cell hematologic tumors | within 3 years after infusion
  OS will be assessed from CAR-T cell infusion to death or last follow-up (censored).
The Peripheral blood vector copy number of patients of CD19&CD22 dual-target CAR-T cell therapy in relapsed/refractory B-cell hematological malignancies | within 3 years after infusion
  Quantity of CD19&CD22 CAR copies in peripheral blood will be determined by using flow cytometry and quantitative polymerase chain reaction.
The Cmax of CAR T cells of CD19&CD22 dual-target CAR-T cell therapy in relapsed/refractory B-cell hematological malignancies | within 3 years after infusion
  The highest concentration of CAR T cells amplified in peripheral blood (Cmax) during the treatment of relapsed/refractory B-cell hematological malignancies
The Tmax of CAR T cells of CD19&CD22 dual-target CAR-T cell therapy in relapsed/refractory B-cell hematological malignancies | within 3 years after infusion
  Time to maximum concentration of CAR T cells in peripheral blood (Tmax) during the treatment of relapsed/refractory B-cell hematological malignancies
The AUC28D of CAR T cells of CD19&CD22 dual-target CAR-T cell therapy in relapsed/refractory B-cell hematological malignancies | within 3 years after infusion
  Area under the curve of peripheral blood CAR T cells at 28 days in peripheral blood (AUC28D) during the treatment of relapsed/refractory B-cell hematological malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, M.D., Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Background] Frank MJ, Baird JH, Kramer AM, Srinagesh HK, Patel S, Brown AK, Oak JS, Younes SF, Natkunam Y, Hamilton MP, Su YJ, Agarwal N, Chinnasamy H, Egeler E, Mavroukakis S, Feldman SA, Sahaf B, Mackall CL, Muffly L, Miklos DB; CARdinal-22 Investigator group. CD22-directed CAR T-cell therapy for large B-cell lymphomas progressing after CD19-directed CAR T-cell therapy: a dose-finding phase 1 study. Lancet. 2024 Jul 27;404(10450):353-363. doi: 10.1016/S0140-6736(24)00746-3. Epub 2024 Jul 9. PMID 38996463
- [Background] Spiegel JY, Patel S, Muffly L, Hossain NM, Oak J, Baird JH, Frank MJ, Shiraz P, Sahaf B, Craig J, Iglesias M, Younes S, Natkunam Y, Ozawa MG, Yang E, Tamaresis J, Chinnasamy H, Ehlinger Z, Reynolds W, Lynn R, Rotiroti MC, Gkitsas N, Arai S, Johnston L, Lowsky R, Majzner RG, Meyer E, Negrin RS, Rezvani AR, Sidana S, Shizuru J, Weng WK, Mullins C, Jacob A, Kirsch I, Bazzano M, Zhou J, Mackay S, Bornheimer SJ, Schultz L, Ramakrishna S, Davis KL, Kong KA, Shah NN, Qin H, Fry T, Feldman S, Mackall CL, Miklos DB. CAR T cells with dual targeting of CD19 and CD22 in adult patients with recurrent or refractory B cell malignancies: a phase 1 trial. Nat Med. 2021 Aug;27(8):1419-1431. doi: 10.1038/s41591-021-01436-0. Epub 2021 Jul 26. PMID 34312556
- [Background] Fry TJ, Shah NN, Orentas RJ, Stetler-Stevenson M, Yuan CM, Ramakrishna S, Wolters P, Martin S, Delbrook C, Yates B, Shalabi H, Fountaine TJ, Shern JF, Majzner RG, Stroncek DF, Sabatino M, Feng Y, Dimitrov DS, Zhang L, Nguyen S, Qin H, Dropulic B, Lee DW, Mackall CL. CD22-targeted CAR T cells induce remission in B-ALL that is naive or resistant to CD19-targeted CAR immunotherapy. Nat Med. 2018 Jan;24(1):20-28. doi: 10.1038/nm.4441. Epub 2017 Nov 20. PMID 29155426
- [Background] Cordoba S, Onuoha S, Thomas S, Pignataro DS, Hough R, Ghorashian S, Vora A, Bonney D, Veys P, Rao K, Lucchini G, Chiesa R, Chu J, Clark L, Fung MM, Smith K, Peticone C, Al-Hajj M, Baldan V, Ferrari M, Srivastava S, Jha R, Arce Vargas F, Duffy K, Day W, Virgo P, Wheeler L, Hancock J, Farzaneh F, Domning S, Zhang Y, Khokhar NZ, Peddareddigari VGR, Wynn R, Pule M, Amrolia PJ. CAR T cells with dual targeting of CD19 and CD22 in pediatric and young adult patients with relapsed or refractory B cell acute lymphoblastic leukemia: a phase 1 trial. Nat Med. 2021 Oct;27(10):1797-1805. doi: 10.1038/s41591-021-01497-1. Epub 2021 Oct 12. PMID 34642489
- [Background] Dual CD19/CD22 CAR T Cells Show Feasibility in Pediatric/Young Adult B-ALL. Cancer Discov. 2021 Dec 1;11(12):2958. doi: 10.1158/2159-8290.CD-RW2021-150. PMID 34686527